CLINICAL TRIAL: NCT01750177
Title: Effect of Sedentary Screen Time Activities Before a Meal on Food Intake in Girls
Brief Title: Sedentary Screen Time Activities on Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Collaborators: Mount Saint Vincent University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Assistant Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: REB 2012-120-002
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Exogenous Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Television Viewing (Experimental): Television viewing before mealtime
  Interventions: Behavioral: Television Viewing before mealtime
- Video Game Playing (Experimental): Video Game Playing before mealtime
  Interventions: Behavioral: Video Game Playing
- Computer Use (Experimental): Computer Use before mealtime
  Interventions: Behavioral: Computer Use
- Sitting Quietly (Experimental): Sitting Quietly before mealtime
  Interventions: Behavioral: Sitting quietly

INTERVENTIONS:
Behavioral: Television Viewing before mealtime
  Arms: Television Viewing
Behavioral: Video Game Playing
  Arms: Video Game Playing
Behavioral: Computer Use
  Arms: Computer Use
Behavioral: Sitting quietly
  Arms: Sitting Quietly

SUMMARY:
The purpose is to investigate the effect of sedentary screen time activities on food intake and subjective appetite in 9- to 14-year old normal weight and overweight/obese girls. The investigators hypothesize that pre-meal exposure to screen time activities for 45 minutes increases subjective appetite and food intake at the next meal. Food intake will be measured immediately following screen-time exposure, and subjective appetite measured throughout the study period at 0, 15, 30, 45 and 75 minutes.

ELIGIBILITY:
Inclusion Criteria:

* healthy girls with no emotional, behavioral or learning problems

Exclusion Criteria:

* boys

Ages: 9 Years to 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Food Intake (kcal) | measured at 45 minutes after the treatment

SECONDARY OUTCOMES:
Subjective appetite | 0-75 minutes
  Subjective appetite (in mm) determined by visual analogue scale

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Department of Applied Human Nutrition, Halifax, Nova Scotia
  - School of Nutrition, Ryerson University, Toronto, Ontario

REFERENCES:
- [Derived] Totosy de Zepetnek JO, Pollard D, Welch JM, Rossiter M, Faghih S, Bellissimo N. Pre-meal screen-time activities increase subjective emotions, but not food intake in young girls. Appetite. 2017 Apr 1;111:32-37. doi: 10.1016/j.appet.2016.12.025. Epub 2016 Dec 21. PMID 28011003